CLINICAL TRIAL: NCT02204176
Title: Exercise Behavior Among Young Adults Study
Acronym: EBYA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Phuong Vo, Graduate Student, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 072613B3F
Record Dates: First submitted 2014-07-25; First posted 2014-07-30 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Exercise info only (Sham Comparator): Participants in the "exercise information only" group will engage in a group discussion with the principal investigator to discuss what constitutes regular physical activity and benefits of exercise and basic tips on the activity itself. Guidelines for prescribing suggested exercises will be based on recommendations from the U.S. Department of Health and Human Services (USDHHS, 2008) as well as risks associated with exercise and how they can be reduced.
  Interventions: Other: Exercise info; Device: pedometer
- Exercise info + implementation intentions (Experimental): Participants in the "exercise information plus implementation intentions" group will engage in a group discussion with the principal investigator to discuss all of the components from the exercise information only approach, but with more emphasis on how to create implementation intentions. Discussions will revolve around possible barriers to exercise plans and how to overcome/address those barriers by making specific plans of when and where to exercise, along with designating which types of exercises they will perform and for how long (or how many repetitions).
  Interventions: Other: Exercise info; Other: Implementation intentions; Device: pedometer
- Exercise info + implementation intentions + industriousness (Experimental): Participants in the "exercise information plus implementation intentions plus industriousness training" group will engage in a group discussion with the principal investigator to discuss all of the components from the second approach as well as include findings linking industriousness and exercise behavior. Participants will be directed to think about and generate solutions to how they can become more industrious and monitor their efforts despite the difficulties they may face and relate these solutions to help them engage in more exercise behavior.
  Interventions: Other: Exercise info; Other: Implementation intentions; Other: Industriousness; Device: pedometer

INTERVENTIONS:
Other: Exercise info — Discussion:
  * benefits of exercise
  * types of exercise
  * exercise guidelines
  * components of an exercise session
  * how to reduce risk of injuries
Other: Implementation intentions — Discussion of:
  * barriers to exercise and how to address/overcome barriers
  * how to create detailed exercise plans
  Arms: Exercise info + implementation intentions; Exercise info + implementation intentions + industriousness
Other: Industriousness — Discussion of:
  * realistic monitoring of efforts related to exercise
  * reaching and pushing past thresholds for sustained effort for exercise
  Arms: Exercise info + implementation intentions + industriousness
Device: pedometer

SUMMARY:
The rate of adult obesity in the United States has increased more than two times since 1970, and the rate of child-teen obesity has increased by four times. One of the antecedents of obesity is an inactive lifestyle. Exercise has been known to be associated with increases in both physical and mental health by increasing longevity, preventing risk of obesity, coronary heart disease, and hypertension, and increasing self-esteem and overall quality of life. The broad aim of the current study is to investigate the effectiveness of psychoeducational training to increase exercise activity initiation and maintenance in young adults.

The goal of this study is to compare three training approaches for college students to increase exercise behavior. One approach provides general information on the different types of exercises and benefits of engaging in exercise behavior after an initial questionnaire assessment session. A second approach includes the general exercise information and questionnaire assessment as well as training on how to create specific goal intentions (i.e., implementation intentions) to aid in exercise initiation. A third approach uses all the components of the second approach but also tests the utility of a personality-informed module by incorporating concepts from the theory of learned industriousness. It is expected that the third approach will be the most effective in helping participants initiate and maintain their exercise activities during the course of the study duration.

DETAILED DESCRIPTION:
The aims of the study (mentioned in the Brief Summary) will be addressed using a 6-month multi-wave assessment of approximately 200 college students. Participants will be randomly assigned to one of the three approaches once it is determined they meet study criteria. Random assignment will occur when the participants are scheduled for the first session.

All participants will partake in three group sessions. The first session will take approximately 2 hours to complete. The second and third sessions will be scheduled 2 and 6 months after the first session and will take approximately 45 minutes each to complete.

In the initial session for the first approach, the group session will include discussion of what constitutes regular physical activity and benefits of exercise and basic tips on the activity itself. Guidelines for prescribing suggested exercises will be based on recommendations from the U.S. Department of Health and Human Services as well as risks associated with exercise and how they can be reduced.

In the initial session for the second approach, the group session will include discussion of all the components from the first approach, but with more emphasis on how to create implementation intentions. Discussions will revolve around possible barriers to exercise plans and how to overcome those barriers by making specific plans of when and where to exercise, along with designating which types of exercises they will perform and for how long (or how many repetitions).

In the initial session for the third approach, the group session will include discussion of all the components from the second approach as well as include findings on industriousness. Participants will be directed to think about and generate solutions to how they can become more industrious despite the difficulties they may face and relate these solutions to help them engage in more exercise behavior.

For all approaches, participants will complete questionnaires regarding aspects of their personality, attitudes regarding exercise, beliefs about the positive and negative effects of exercise, confidence in engaging in exercise despite barriers, and current levels of exercise. Participants' body mass index will also be measured. All participants will be given an exercise booklet tailored to their respective approaches to record their exercise behavior during the three weeks following the initial session. They will also be loaned a pedometer that will be used to track their overall daily activities for the same three-week period. Participants in the third approach will also receive booster contacts (to encourage them to think about their efforts and monitoring of physical activity) every two weeks starting after the three-week tracking period until their six-month follow up (total of 11 booster contacts).

The first session will be video and audio recorded to check on and ensure presentation consistency. At the end of the first session, participants will be given a post-session survey to gauge how well materials were presented and to determine how much information participants felt they gained from the session. When participants return their daily exercise diaries and pedometers, they will also complete a condensed set of measures (similar to those in the first session) to track any changes experienced during the three-week tracking period.

For the 2- and 6-month follow-up sessions, participants in all approaches will complete the same questionnaires as in the initial session and have their body mass index measured.

Power analyses conducted via G*Power, 3.1.6 indicated that 159 participants will be needed to detect an effect size of F of 0.25 with alpha error probability at 0.05 and power at 1-Β =.80. Oversampling by 25% will occur to account for possible attrition from the study, thereby making the target N = 200.

ELIGIBILITY:
Inclusion Criteria:

* be currently enrolled in full-time university coursework
* be between 18 and 24 years old
* understand and respond to screening questions in English
* be able to read at a Grade 6 level
* have adequate health, as assessed by having a body mass index between 18.5 and 29.9 (anyone with a BMI of 30+ is considered obese; National Heart, Lung, & Blood Institute, 2012) to ensure that regular, moderate to intense exercise activity will not negatively affect health
* identify as individuals who have tried to initiate and continue an exercise regimen sometime in the past but have been unable to maintain the activity
* indicate the desire to initiate physical activity at the current time
* be willing to attempt to maintain an exercise schedule during the three-week intervention period to which they will be randomly assigned
* be willing to participate in the 2-month and 6-month follow up periods

Exclusion Criteria:

* not already be meeting current USDHHS physical activity recommendations (i.e., at least 150 minutes of moderate-intensity exercise per week)
* not have major cognitive impairments (i.e., assessed by whether they can understand and respond adequately to all screening questions)
* not report consuming more than three (women) or four (men) alcoholic drinks per day (as this may interfere with their ability to engage in physical activity and confound study results)
* not be pregnant
* not have children
* not have preexisting physical limitations or recent injuries
* not have major cognitive impairments (i.e., assessed by whether they can understand and respond adequately to all screening questions)

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phuong T Vo, BA, Principal Investigator — Wayne State University; Tim D Bogg, PhD, Study Director — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Eisenberger R. Learned industriousness. Psychol Rev. 1992 Apr;99(2):248-67. doi: 10.1037/0033-295x.99.2.248. PMID 1594725
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] McAuley E & Rudolph D. Physical activity, aging, and psychological well-being. Journal of Aging and Physical Activity 3: 67-96, 1995.
- [Background] National Heart, Lung, and Blood Institute. (2012, July 13). How are overweight and obesity diagnosed? Retrieved from http://www.nhlbi.nih.gov/health/health-topics/topics/obe/diagnosis.html
- [Background] U.S. Department of Health and Human Services. 2008 physical activity guidelines for Americans. Washington DC: U.S. Department of Health and Human Services, 2008.
- [Background] Webb TL & Sheeran P. Identifying good opportunities to act: Implementation intentions and cue discrimination. European Journal of Social Psychology, 34: 407-419, 2004.
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Benosovich SV, Rossi JS, Norman GJ, & Nigg CR. Development of a multidimensional measure of exercise self-efficacy. Annals of Behavioral Medicine, 20: S190, 1998.
- [Background] Roberts BW, Bogg T, Walton KE, Chernyshenko OS, & Stark. A lexical investigation of the lower-order structure of conscientiousness. Journal of Research in Personality, 38: 164-178, 2004.
- [Background] Hill PL, Roberts BW. The role of adherence in the relationship between conscientiousness and perceived health. Health Psychol. 2011 Nov;30(6):797-804. doi: 10.1037/a0023860. Epub 2011 May 23. PMID 21604876

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise Information: This group was presented with information that defined and described regular exercise, its benefits, and guidance for using proper form in exercise to minimize the risk of injury. Guidelines for prescribing suggested physical activities were based on recommendations from the USDHHS (2008). These sessions lasted ~90 minutes.
- Action Planning: This group discussed all the components from the session for the information-only group with an additional emphasis on how to create action plans. Discussions revolved around possible ways and times of the day to engage in exercise by making specific action plans that designate when, where, and how. Participants were shown how to create an example action plan and guided in writing their own exercise action plans for as many days as they desired in the three-week tracking period in their exercise booklets. Emphasis was placed on the specificity and feasibility of the plans. These sessions lasted ~120 minutes.
- Realistic Effort Action Planning: This group discussed all components from the action planning condition. Discussion in this group also emphasized the importance of persistence and effortful control in daily life and how these attributes can be transferred to exercise plans. Participants were encouraged to identify their threshold for exerting effort toward exercise based on past experiences and applying that awareness to their planned exercises. They were guided in creating action plans that considered not only past external barriers (e.g., schedule, fitness level, and environment) but also previous internal barriers (i.e., resistance and/or aversiveness to physical exertion) and create plans that would help them avoid repeating the same circumstances. Participants were also asked to realistically consider how much past exercise they have previously engaged in and to refine those estimates to serve as starting points for subsequent small increases in planned exercise. These group sessions lasted ~120 minutes.
Period: Overall Study
Arm/Group | Exercise Information | Action Planning | Realistic Effort Action Planning
Started | 74 | 73 | 74
Completed | 64 | 61 | 58
Not Completed | 10 | 12 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Information | Action Planning | Realistic Effort Action Planning | Total
Number analyzed (Participants) | 74 | 73 | 74 | 221
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.39 (1.91) | 20.59 (2.05) | 20.70 (2.18) | 20.56 (2.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 42 | 44 | 132
  Male | 28 | 31 | 30 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 19 | 20 | 15 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 10 | 8 | 29
  White | 34 | 28 | 43 | 105
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 15 | 8 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 74 | 73 | 74 | 221
Strenuous Exercise [Mean (Standard Deviation); unit: times per week] — The Godin Leisure-Time Exercise Questionnaire (GLTEQ; Godin & Shephard, 1985) was used to assess the frequency of typical weekly strenuous, moderate, and mild exercise (open-ended format). Total exercise scores were also computed by multiplying each reported exercise frequency by its metabolic equivalent (MET) and then summing the totals: (strenuous x 9) + (moderate x 5) + (mild x 2) (Godin, Jobin, & Boullon, 1986). Higher scores indicate greater exercise engagement.
  times per week | 1.36 (.17) | 1.44 (.18) | 1.17 (.16) | 1.32 (.10)
Moderate Exercise [Mean (Standard Deviation); unit: times per week] — The Godin Leisure-Time Exercise Questionnaire (GLTEQ; Godin & Shephard, 1985) was used to assess the frequency of typical weekly strenuous, moderate, and mild exercise (open-ended format). Total exercise scores were also computed by multiplying each reported exercise frequency by its metabolic equivalent (MET) and then summing the totals: (strenuous x 9) + (moderate x 5) + (mild x 2) (Godin, Jobin, & Boullon, 1986). Higher scores indicate greater exercise engagement.
  times per week | 1.69 (.17) | 2.40 (.23) | 1.93 (.21) | 2.00 (.12)
Mild Exercise [Mean (Standard Deviation); unit: times per week] — The Godin Leisure-Time Exercise Questionnaire (GLTEQ; Godin & Shephard, 1985) was used to assess the frequency of typical weekly strenuous, moderate, and mild exercise (open-ended format). Total exercise scores were also computed by multiplying each reported exercise frequency by its metabolic equivalent (MET) and then summing the totals: (strenuous x 9) + (moderate x 5) + (mild x 2) (Godin, Jobin, & Boullon, 1986). Higher scores indicate greater exercise engagement.
  times per week | 2.54 (.33) | 2.95 (.34) | 3.03 (.29) | 2.84 (.19)
Total Exercise [Mean (Standard Deviation); unit: total metabolic equivalent] — The Godin Leisure-Time Exercise Questionnaire (GLTEQ; Godin & Shephard, 1985) was used to assess the frequency of typical weekly strenuous, moderate, and mild exercise (open-ended format). Total exercise scores were also computed by multiplying each reported exercise frequency by its metabolic equivalent (MET) and then summing the totals: (strenuous x 9) + (moderate x 5) + (mild x 2) (Godin, Jobin, & Boullon, 1986). Higher scores indicate greater exercise engagement.
  total metabolic equivalent | 28.29 (2.48) | 33.79 (2.87) | 29.23 (2.41) | 30.42 (1.50)
Industriousness [Mean (Standard Deviation); unit: 1(disagree strongly)-5(agree strongly)] — Industriousness was assessed using a 10-item Industriousness scale (Chernyshenko, 2003). Participants rated themselves on a 5-point Likert scale (1 = Disagree strongly, 5 = Agree strongly) indicating the extent to which, for example, they are someone who "has high standards and works toward them; setting goals and achieving them is not very important to me [reversed], [or] invests little effort into my work [reversed] ". Higher scores indicate greater industriousness level.
  1(disagree strongly)-5(agree strongly) | 4.02 (.07) | 4.09 (.07) | 3.89 (.08) | 4.00 (.04)

OUTCOME MEASURES:

1. Primary Outcome: Total Physical Activity
Description: The Godin Leisure-Time Exercise Questionnaire (GLTEQ; Godin & Shephard, 1985) was used to assess the frequency of typical weekly strenuous, moderate, and mild exercise (open-ended format). Total exercise scores were also computed by multiplying each reported exercise frequency by its metabolic equivalent (MET) and then summing the totals: (strenuous x 9) + (moderate x 5) + (mild x 2) (Godin, Jobin, & Boullon, 1986). Higher scores on this scale indicates more exercise engagement.
  Also, participants were loaned a pedometer to obtain objective measures of exercise activity. The pedometers allow participants to enter their weight and height and measure steps taken throughout the day based on this information. The devices automatically reset at midnight and store the information for 30 days.
Time Frame: 2-3 months after initial intervention session
Measure: Mean (Standard Error); unit: total metabolic equivalent
Arm/Group | Exercise Information | Action Planning | Realistic Effort Action Planning
Number analyzed (Participants) | 74 | 73 | 74
total metabolic equivalent | 34.21 (2.59) | 37.80 (2.80) | 39.42 (2.73)

2. Primary Outcome: Total Physical Activity
Description: The Godin Leisure-Time Exercise Questionnaire (GLTEQ; Godin & Shephard, 1985) was used to assess the frequency of typical weekly strenuous, moderate, and mild exercise (open-ended format). Total exercise scores were also computed by multiplying each reported exercise frequency by its metabolic equivalent (MET) and then summing the totals: (strenuous x 9) + (moderate x 5) + (mild x 2) (Godin, Jobin, & Boullon, 1986). Higher scores indicate more exercise engagement.
  Also, participants were loaned a pedometer to obtain objective measures of exercise activity. The pedometers allow participants to enter their weight and height and measure steps taken throughout the day based on this information. The devices automatically reset at midnight and store the information for 30 days.
Time Frame: 6 months after initial intervention session
Measure: Mean (Standard Error); unit: total metabolic equivalent
Arm/Group | Exercise Information | Action Planning | Realistic Effort Action Planning
Number analyzed (Participants) | 74 | 73 | 74
total metabolic equivalent | 38.65 (3.09) | 40.64 (2.43) | 42.39 (2.97)

3. Secondary Outcome: Exercise Self-efficacy
Description: The 18-item multidimensional exercise self-efficacy scale (Benisovich, Rossi, Norman, & Nigg, 1998) assessed participants' confidence in being able to exercise despite bad weather, inconvenience, negative affect, exercising alone, excuse making, and resistance from others. Participants were asked to rate "how confident [they] are to exercise when other things get in the way" on a 5-point Likert scale (1 = Not at all confident, 5 = Extremely confident). Example items include, "I don't have access to exercise equipment," "I don't feel like it," and "I am spending time with friends or family who do not exercise." All items on the scale were averaged for each participant. Higher scores indicate greater self-efficacy for exercise.
Time Frame: 2-3 months after initial intervention session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Exercise Information | Action Planning | Realistic Effort Action Planning
Number analyzed (Participants) | 74 | 73 | 74
units on a scale | 2.92 (.09) | 3.05 (.11) | 3.09 (.10)

4. Secondary Outcome: Exercise Self-efficacy
Description: The 18-item multidimensional exercise self-efficacy scale (Benisovich, Rossi, Norman, & Nigg, 1998) assessed participants' confidence in being able to exercise despite bad weather, inconvenience, negative affect, exercising alone, excuse making, and resistance from others. Participants were asked to rate "how confident [they] are to exercise when other things get in the way" on a 5-point Likert scale (1 = Not at all confident, 5 = Extremely confident; αs = .89-.91 across assessments). Example items include, "I don't have access to exercise equipment," "I don't feel like it," and "I am spending time with friends or family who do not exercise." All items on the scale were averaged for each participant. Higher scores indicate greater self-efficacy.
Time Frame: 6 months after initial intervention session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Exercise Information | Action Planning | Realistic Effort Action Planning
Number analyzed (Participants) | 74 | 73 | 74
units on a scale | 2.95 (.12) | 2.94 (.09) | 3.08 (.11)

5. Other Pre Specified Outcome: Industriousness Level
Description: Industriousness was assessed using a 10-item Industriousness scale (Chernyshenko, 2003). Participants rated themselves on a 5-point Likert scale (1 = Disagree strongly, 5 = Agree strongly) indicating the extent to which, for example, they are someone who "has high standards and works toward them; setting goals and achieving them is not very important to me [reversed], [or] invests little effort into my work [reversed] ". Higher scores indicate greater industriousness level.
Time Frame: 2-3 months after initial intervention session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Exercise Information | Action Planning | Realistic Effort Action Planning
Number analyzed (Participants) | 74 | 73 | 74
units on a scale | 4.01 (.13) | 3.96 (.26) | 3.98 (.25)

6. Other Pre Specified Outcome: Industriousness Level
Description: as for outcome 5
Time Frame: 6 months after initial intervention session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Exercise Information | Action Planning | Realistic Effort Action Planning
Number analyzed (Participants) | 74 | 73 | 74
units on a scale | 4.01 (.09) | 4.07 (.08) | 3.95 (.10)

ADVERSE EVENTS:
Time Frame: 1 year and 5 months
Description: No adverse events occurred during the completion of the present study.
Arm/Group | Exercise Information | Action Planning | Realistic Effort Action Planning
All-Cause Mortality (participants affected / at risk) | 0/221 | 0/221 | 0/221
Serious Adverse Events (participants affected / at risk) | 0/221 | 0/221 | 0/221
Other Adverse Events (participants affected / at risk) | 0/221 | 0/221 | 0/221

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No